CLINICAL TRIAL: NCT01568307
Title: Interactions Between The Serotonin Transporter And Sympathetic Nervous System Activation In Patients With Major Depressive Disorder - Understanding The Link Between The Brain And The Heart
Brief Title: Major Depressive Disorder - Understanding The Link Between The Brain And The Heart
Acronym: MDD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: The Alfred (Other); Monash Medical Centre (Other); Ballarat Health Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 74/12; 1022791 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2012-03-25; First posted 2012-04-02 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2018-11

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Serotonin transporter; Sympathetic nervous system activation; Cardiovascular risk factors; Serotonin re-uptake inhibitor
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Antidepressive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Participants will be prescribed an approved selective serotonin re-uptake inhibitor (SSRI) antidepressant. — The choice of SSRI will be based on clinical judgement and prescribed in line with standard dosing approved by the Therapeutic Goods Administration (TGA).

SUMMARY:
There is strong evidence that patients with major depressive disorder (MDD) have an increased risk of developing coronary heart disease (CHD). This elevated risk is independent of standard risk factors such as smoking, obesity, high cholesterol, diabetes, and high blood pressure. The relative risk of developing CHD is proportional to the severity of depression (the more severe the depression, the more likely the development of CHD).

The sympathetic nervous system (the part of your nervous system that makes your heart beat harder and faster) is responsible for our "flight and fight" response to a threatening situation. It has been determined that increased sympathetic nervous system activation occurs in approximately one in three untreated patients with MDD (with no underlying CHD). There is growing evidence linking elevated sympathetic activity to early stages of kidney dysfunction and an increased incidence of cardiovascular (heart and blood vessel) disease development (eg, heart attacks). Sympathetic nervous system activation over a prolonged period of time may also be associated with abnormal blood pressure regulation and the development of insulin resistance (an important feature of type 2 diabetes).

It has been suggested that a certain gene, known as the serotonin transporter (5-HTT) gene, may be involved. In particular, work from our group indicates that a particular type of this gene, the short form (or "short" allele) may be important in linking MDD, sympathetic nervous activation, and increased cardiac risk.

This study aims to examine the role of the 5-HTT gene on cardiovascular risk factors associated with elevated sympathetic activity in patients with MDD. Additionally, the study will examine the effect of serotonin re-uptake inhibitor (SSRI) therapy on these parameters.

A clearer understanding of these systems and processes will allow for identification of patients with increased cardiac risk and development of risk reduction strategies. Such information is clinically significant given the link between cardiovascular disease and MDD.

Hypothesis 1: That MDD patients carrying the s allele of the 5-HTT transporter have higher sympathetic activity than homozygous ll patients.

Hypothesis 2: that MDD patients with elevated sympathetic activity display early signs of left ventricular hypertrophy (LVH) and diastolic dysfunction.

Hypothesis 3: That MDD patients with high sympathetic activity have greater morning surges in blood pressure than patients with normal sympathetic activity.

Hypothesis 4: That MDD patients with elevated sympathetic activity display early signs of insulin resistance.

Hypothesis 5: That SSRI therapy, in particular in those who carry the s allele of the 5-HTT, has a favourable effect on blood pressure variability and morning surge in blood pressure, sympathetic stress reactivity, and markers of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years.
* Capable of understanding and willing to provide signed and dated written, voluntary informed consent in advance of any protocol-specific procedures.
* MDD or MDD with melancholia according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria. Patients with comorbid panic or anxiety disorders will be included if MDD is the primary diagnosis.
* Hamilton Depression (HAM D) > 18.
* Beck Depression Inventory (BDI-II) > 18.

Exclusion Criteria:

* Aged < 18 or > 70 years.
* Current antidepressant treatment.
* Previous failed response to SSRI treatment at the maximum tolerated dose for at least 4 weeks.
* Known or suspected hypersensitivity to the prescribed antidepressant or any of its ingredients.
* Current high suicide risk.
* Comorbid panic or anxiety disorders as the primary diagnosis.
* Pre-existing and/or current diagnosed heart disease.
* Comorbid medical conditions including type 1 diabetes, medicated hypertension, epilepsy, bleeding disorders, alcohol/drug dependence, infectious blood diseases, psychotic disorders, personality disorders, eating disorders, mental retardation, dementia (ie, Mini Mental State Examination [MMSE] < 23), or gastrointestinal illness or previous bariatric (weight loss) surgery that may impair antidepressant absorption.
* Clinically significant abnormalities on examination or laboratory testing and clinically significant medical conditions not listed above that are serious and/or unstable.
* Pregnant or breastfeeding women.
* Women of childbearing potential (WOCP) who are not using medically accepted contraception (ie, intrauterine devices [IUDs], hormonal contraceptives [oral, depot, patch or injectable], and double barrier methods such as condoms or diaphragms with spermicidal gel or foam). Women who are postmenopausal (amenorrhea for at least 12 consecutive months) or surgically sterile are not considered to be WOCP.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-05; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Proportion of MDD patients carrying the s allele of the 5-HTT transporter that have higher sympathetic activity than homozygous ll patients. | up to 12 weeks
  Participants will be prescribed an approved SSRI in line with standard practice.The investigators will explore the association between the degree of sympathetic nervous activation and 5-HTT genotype in patients with MDD. They do not plan to examine the role of the 5-HTT genotype on MDD development. They will examine the relationship between the degree of sympathetic nervous system activity and early signs of cardiac structure and function abnormalities, insulin resistance, and morning surge in blood pressure. This may help in identifying MDD patients who are at an increased risk.

SECONDARY OUTCOMES:
To determine the association between sympathetic activity and left ventricular hypertrophy. | Baseline
  The investigators will measure the relationship between sympathetic nervous activity and left ventricular mass in patients with MDD. ECG, ECHO, and blood pressure data will be used to test the hypothesis that MDD patients with elevated sympathetic activity display early signs of LVH and diastolic dysfunction.
Change from baseline in the magnitude of morning surge in blood pressure. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between sympathetic nervous system activity and stress reactivity to the morning surge in blood pressure in patients with MDD. Blood pressure data will be used to test the hypothesis that MDD patients with high sympathetic activity have greater morning surges in blood pressure than patients with normal sympathetic activity.
Change from baseline in insulin resistance. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between sympathetic nervous activity and stress reactivity to signs of insulin resistance in patients with MDD. Oral glucose tolerance test data will be used to test the hypothesis that MDD patients with elevated sympathetic activity display early signs of insulin resistance.
Change from baseline on markers of cardiac risk. | Baseline and following 12 weeks of antidepressant treatment.
  The investigators will explore the association between SSRI therapy and markers of cardiac risk. They will test the hypothesis that SSRI therapy, in particular in those who carry th s allele of the 5-HTT, has a favourable effect on blood pressure variability and morning surge in blood pressure, sympathetic stress reactivity, and markers of insulin resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Lambert, Study Director — Baker IDI Heart & Diabetes Institute; David Barton, Principal Investigator — Monash Medical Centre; Abdul Khalid, Principal Investigator — Ballarat Health Services
Locations (4):
- Australia (4):
  - Ballarat Health Service Psychiatric Services, Ballarat, Victoria
  - Monash Medical Centre - Monash Health, Clayton, Victoria
  - Alfred and Baker Medical Unit - Alfred Hospital, Melbourne, Victoria
  - Baker IDI Heart & Diabetes Institute, Melbourne, Victoria